CLINICAL TRIAL: NCT01209221
Title: A Phase 1 Placebo-controlled, Randomized, Observer-blind Combined Single and Multiple Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO5271983 in Healthy Subjects.
Brief Title: A Single Ascending And Multiple Ascending Dose Study of RO5271983 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NP25342
Record Dates: First submitted 2010-09-24; First posted 2010-09-27 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: RO5271983 - SAD
- 2 (Experimental)
  Interventions: Drug: RO5271983 - MAD
- 3 (Placebo Comparator)
  Interventions: Drug: Placebo - SAD
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo - MAD

INTERVENTIONS:
Drug: Placebo - MAD — Once or twice daily doses of matching placebo to RO5271983 for 14 days
  Arms: 4
Drug: Placebo - SAD — Single dose of matching placebo to RO5271983 for up to 3 periods
  Arms: 3
Drug: RO5271983 - MAD — Once or twice daily doses of RO5271983 for 14 days
  Arms: 2
Drug: RO5271983 - SAD — Single dose of RO5271983 at each period (for up to 3 periods)
  Arms: 1

SUMMARY:
This placebo-controlled, randomized, observer-blind, dose-ascending study will investigate the safety, tolerability, pharmacokinetics and pharmacodynamics of single and multiple doses of RO5271983 in healthy volunteers. Healthy volunteers will be randomized to receive either a single oral dose of RO5271983 or placebo in the SAD part or multiple oral doses of RO5271983 or placebo in the MAD part. The anticipated time on study treatment is approximately 14 weeks for the SAD part and up to 8 weeks for the MAD part.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, 18-65 years of age
* Body Mass Index (BMI) between 18 and 32 kg/m2, inclusive
* In the SAD, females subjects must be surgically sterile or post-menopausal for the past year; in the MAD females may be of child-bearing potential but must use 2 methods of highly effective contraception

Exclusion Criteria:

* A history of clinically relevant cardiovascular, gastrointestinal, hepatic, renal, endocrine, pulmonary, neurological, psychiatric, allergic or skin disease
* Clinical significant abnormalities in laboratory test results
* Symptoms of an infectious disease including upper respiratory tract infection within one month of study start or a history of recurrent infections
* Smokers of >5 cigarettes/day within 3 months prior to admission and unable to stop smoking during study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2010-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Single ascending dose (SAD): Pharmacokinetics (plasma concentration) of RO5271983 | up to 240 hours
Single ascending dose (SAD): Safety (incidence of adverse events) | 14 weeks
Single ascending dose (SAD): Tolerability (e.g. vital signs) | 14 weeks
Multiple ascending doses (MAD): Pharmacokinetics (plasma concentration) of RO5271983 | 17 days
Multiple ascending doses (MAD): Safety (incidence of adverse events) | 8 weeks
Multiple ascending doses (MAD): Tolerability (e.g. vital signs) | 8 weeks

SECONDARY OUTCOMES:
Effect of food on pharmacokinetics of RO5271983 | up to 240 hours
Single ascending dose (SAD): Pharmacodynamics (blood analysis) of RO5271983 | 72 hours
Multiple ascending doses (MAD): Pharmacodynamics (blood analysis) of RO5271983 | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Christchurch, New Zealand